CLINICAL TRIAL: NCT01556815
Title: Phase II Trail of Sorafenib Combined With Transarterial Chemoembolization in HBV-infected Patients With Intermediate Hepatocellular Carcinoma
Brief Title: Sorafenib Combined With Transarterial Chemoembolization in Treating HBV-infected Patients With Intermediate Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinlong Song, Chief, Division of Interventional Therapy, Shandong Cancer Hospital and Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShandongCHI-001
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: PHENYTOIN/SORAFENIB [VA Drug Interaction]; Liver Neoplasms; Carcinoma, Hepatocellular; Digestive System Neoplasms; Neoplasms by Site; Liver Diseases; Adenocarcinoma; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; DOXORUBICIN/TRASTUZUMAB [VA Drug Interaction]; HBV
Keywords: Hepatocellular Carcinoma; Sorafenib; Transarterial Chemoembolization; HBV
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular; Digestive System Neoplasms; Neoplasms by Site; Liver Diseases; Adenocarcinoma; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group TACE (Active Comparator): Patients who undergo TACE
  Interventions: Procedure: Transarterial Chemoembolization (TACE)
- Group Combination (Experimental): Patients who are treated with sorafenib combined with TACE
  Interventions: Other: Sorafenib in combination with TACE

INTERVENTIONS:
Procedure: Transarterial Chemoembolization (TACE) — Procedure:TACE TACE will be carried out with an emulsion of 50mg doxorubicin with lipiodol in a total volume of 10-20 mL; additional embolisation will be carried out with gelatin sponge particles. TACE will be repeated every 4 weeks for 2 cycles; additional cycles will be offered if clinically indicated .
  Arms: Group TACE
Other: Sorafenib in combination with TACE — Drug: Sorafenib All patients will receive Sorafenib (800 mg/day) p.o. beginning one week after the first TACE and every day thereafter until patient death or premature withdrawal from study.
  Procedure: TACE
  TACE will be carried out with an emulsion of 50mg doxorubicin with lipiodol in a total volume of 10-20 mL; additional embolisation will be carried out with gelatin sponge particles. TACE will be repeated every 4 weeks for 2 cycles; additional cycles will be offered if clinically indicated .
  Other Names: Sorafenib:Nexavar(brand name)
  Arms: Group Combination

SUMMARY:
Transarterial chemoembolization (TACE) is widely used for unresectable hepatocellular carcinoma (HCC). However, the hypoxia caused by TACE in surviving tumor cell leads to release of angiogenic and growth factors contributing to poor outcome. Sorafenib can block tumor cell proliferation and angiogenesis. The hypothesis is that patients with unresectable HCC may benefit from sorafenib in combination with TACE.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed as HCC according to European Association for Study of the Liver criteria.
* BCLC stage B
* Child-Pugh class A
* ECOG performance status of 0
* Etiology: Hepatitis B virus(HBV) infection
* Written informed consent (approved by the Institutional Review Board [IRB]obtained prior to any study specific screening procedures
* Patient must be able to comply with the protocol
* Age 18-80 years
* Haematology:Absolute neutrophil count (ANC) > 1 x 109/L, Platelet count > 40 x 109/L, Haemoglobin > 9 g/dL (may be transfused to maintain or exceed this level) Prothrombin time international normalized ratio < 1.5
* Biochemistry:Total bilirubin < 2 mg/dL Serum creatinine < 1.5 x the upper limit of normal
* Life expectancy of > 3 months

Exclusion Criteria:

* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 5 x the upper limit of normal
* Other severe concomitant disease that may reduce life expectancy
* uncontrolled hypertension
* Pregnancy (positive serum pregnancy test) or lactation
* Uncontrolled hypertension
* Serious, non-healing wound, ulcer, or bone fracture
* Currently or recent (within the 30 days prior to starting study treatment) treatment of another investigational drug or participation in another investigational study
* Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents ( ≤ 6 months prior to study entry), myocardial infarction ( ≤ 6 months prior to study entry), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication
* Evidence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of Sorafenib/TACE or patient at high risk from treatment complications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of sorafenib in increasing the effectiveness of transarterial chemoembolization (TACE) | 1 year
  Measure:time-to-proression

SECONDARY OUTCOMES:
safety of sorafenib in combination with TACE | 6 months
  Measure: incidence and grade of adverse events in patients treated with sorafenib combined with TACE (group B)
Survival in the two treatment groups | 2 years
  Measured from the date of TACE until the date of death or last visit

CONTACTS AND LOCATIONS:
Overall Officials: Jinlong Song, MD, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China